CLINICAL TRIAL: NCT06209632
Title: Effects of Mirror Therapy Combined With Contralaterally Controlled Functional Electrical Stimulation on Functional Recovery and Neuroplasticity in Patients With Peripheral Nerve Injury
Brief Title: Mirror Therapy Combined With Contralaterally Controlled Functional Electrical Stimulation for Peripheral Nerve Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 202309076RINA
Record Dates: First submitted 2024-01-03; First posted 2024-01-17 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Peripheral Nerve Injury
Keywords: mirror therapy; electrical stimulation; neuroplasticity; peripheral nerve injury
MeSH Terms: conditions — Peripheral Nerve Injuries | interventions — Mirror Movement Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- MT and CCFES group (Experimental): mirror therapy combined with contralaterally controlled functional electrical stimulation to perform hand exercises
  Interventions: Behavioral: mirror therapy; Device: contralaterally controlled functional electrical stimulation; Behavioral: conventional physiotherapy
- Sham MT and CCFES group (Sham Comparator): sham mirror therapy with contralaterally controlled functional electrical stimulation to perform hand exercises
  Interventions: Device: contralaterally controlled functional electrical stimulation; Behavioral: conventional physiotherapy
- Control group (Active Comparator): conventional physiotherapy
  Interventions: Behavioral: conventional physiotherapy

INTERVENTIONS:
Behavioral: mirror therapy — 30 minutes of intervention, twice a week, and a total of 12 weeks
  Arms: MT and CCFES group
Device: contralaterally controlled functional electrical stimulation — 30 minutes of intervention, twice a week, and a total of 12 weeks
  Arms: MT and CCFES group; Sham MT and CCFES group
Behavioral: conventional physiotherapy — 50 minutes of intervention, twice a week, and a total of 12 weeks

SUMMARY:
The goal of this trial is to evaluate the effects of mirror therapy combined with contralaterally controlled functional electrical stimulation on motor recovery and neuroplasticity in patients with peripheral nerve injury. The main questions it aims to answer are Question 1: To compare corticomuscular coherence between the groups of mirror therapy combined with contralaterally controlled functional electrical stimulation, sham mirror therapy combined with contralaterally controlled functional electrical stimulation, and control group.

Question 2: To compare sensorimotor recovery between the groups of mirror therapy combined with contralaterally controlled functional electrical stimulation, sham mirror therapy combined with contralaterally controlled functional electrical stimulation, and control group.

Question 3: To evaluate the effects of each intervention on corticomuscular coherence and sensorimotor recovery 12 weeks post-intervention.

Participants will be asked to exercise their affected hand together with the unaffected hand while receiving contralaterally controlled electrical stimulation in front of the mirror or sham mirror. Researchers will compare the effects of mirror therapy combined with contralaterally controlled functional electrical stimulation on corticomuscular coherence and sensorimotor recovery with the other groups.

DETAILED DESCRIPTION:
The goal of this trial is to evaluate the effects of mirror therapy combined with contralaterally controlled functional electrical stimulation on motor recovery and neuroplasticity in patients with peripheral nerve injury. The main questions it aims to answer are:

Question 1: To compare corticomuscular coherence between the groups of mirror therapy combined with contralaterally controlled functional electrical stimulation, sham mirror therapy combined with contralaterally controlled functional electrical stimulation, and control group.

Question 2: To compare sensorimotor recovery between the groups of mirror therapy combined with contralaterally controlled functional electrical stimulation, sham mirror therapy combined with contralaterally controlled functional electrical stimulation, and control group.

Question 3: To evaluate the effects of each intervention on corticomuscular coherence and sensorimotor recovery 12 weeks post-intervention.

Eligible participants will be randomized into three groups:

MT and CCFES group: mirror therapy combined with contralaterally controlled functional electrical stimulation Sham MT and CCFES group: Sham mirror therapy combined with contralaterally controlled functional electrical stimulation Control group: conventional physiotherapy.

Each participant will receive conventional physiotherapy for 50 minutes daily, twice a week for 12 weeks. Conventional physiotherapy includes scar management, joint range of motion exercise, strengthening, stretching, and functional training. Participants in the MT and CCFES group or Sham MT and CCFES group will receive 30 minutes daily, twice a week of the intervention for 12 weeks in addition to the conventional physiotherapy. In the MT and CCFES group, the participants will sit in front of the mirror and watch the mirror reflection of the unaffected hands. At the same time, contralaterally controlled electrical stimulation will be conducted to make the affected hands move with the unaffected hands. The participants in the Sham MT and CCFES group will sit in front of the mirror without mirror reflection, but doing the exercise with contralaterally controlled functional electrical stimulation. All participants will receive the evaluations at baseline and 12 weeks after the intervention. The evaluations include:

Electroencephalography of α and β bands from the sensorimotor cortices will be recorded.

Electromyography will be performed during maximum isometric pinch or lateral pinch strength measurements.

Maximum isometric grip strength, tip pinch strength, lateral pinch strength, sensation tests, and upper extremity function will be measured.

ELIGIBILITY:
Inclusion Criteria:

* newly diagnosed median or ulnar nerve transection injury of the forearm in the past 6 months
* sufficient communication in the Chinese language
* being able to follow instructions
* the presence of target muscle denervation (e.g. muscle atrophy, inability to actively contract)
* less than 10% surface EMG activity during pinch evaluation compared to the unaffected side

Exclusion Criteria:

* had central nervous disease
* had a recent (1 year) history of nerve entrapment syndrome
* had a history of latent neuropathy, such as diabetes or dialysis

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2024-03-29 (Actual); Primary Completion 2025-11-30 (Actual); Study Completion 2025-11-30 (Actual)

PRIMARY OUTCOMES:
change from baseline in corticomuscular coherence at week 12 | baseline, week 12
  coherence will be used to analyze the interaction between the electroencephalogram activation and electromyography activation

SECONDARY OUTCOMES:
change from baseline in grip strength at week 12 | baseline, week 12
  average grip strength measured for 3 times in killograms
change from baseline in pinch strength at week 12 | baseline, week 12
  average lateral pinch and palmar pinch measured for 3 times in killograms
change from baseline in sensation on Semmes-Weinstein monofilament test at week 12 | baseline, week 12
  force in grams
change from baseline in function on Disabilities of the Arm, Shoulder, and Hand outcome questionnaire at week 12 | baseline, week 12
  A total scale from 1 to 100. Higher scores indicate greater disability.
change from baseline in maximum voluntary isometric contraction in surface EMG at week 12 | baseline, week 12
  muscle activities of target muscles measured during pinch strength for 3 times in percentage

CONTACTS AND LOCATIONS:
Overall Officials: Yueh-Hsia Chen, PhD, Principal Investigator — National Taiwan University, School of Medicine
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rizzo M, Petrini L, Del Percio C, Lopez S, Arendt-Nielsen L, Babiloni C. Mirror visual feedback during unilateral finger movements is related to the desynchronization of cortical electroencephalographic somatomotor alpha rhythms. Psychophysiology. 2022 Dec;59(12):e14116. doi: 10.1111/psyp.14116. Epub 2022 Jun 3. PMID 35657095
- [Background] Bello UM, Kranz GS, Winser SJ, Chan CCH. Neural Processes Underlying Mirror-Induced Visual Illusion: An Activation Likelihood Estimation Meta-Analysis. Front Hum Neurosci. 2020 Jul 31;14:276. doi: 10.3389/fnhum.2020.00276. eCollection 2020. PMID 32848663
- [Background] Deconinck FJ, Smorenburg AR, Benham A, Ledebt A, Feltham MG, Savelsbergh GJ. Reflections on mirror therapy: a systematic review of the effect of mirror visual feedback on the brain. Neurorehabil Neural Repair. 2015 May;29(4):349-61. doi: 10.1177/1545968314546134. Epub 2014 Aug 26. PMID 25160567
- [Background] Cengiz B, Vuralli D, Zinnuroglu M, Bayer G, Golmohammadzadeh H, Gunendi Z, Turgut AE, Irfanoglu B, Arikan KB. Analysis of mirror neuron system activation during action observation alone and action observation with motor imagery tasks. Exp Brain Res. 2018 Feb;236(2):497-503. doi: 10.1007/s00221-017-5147-5. Epub 2017 Dec 11. PMID 29230518
- [Background] Zhang JJQ, Fong KNK, Welage N, Liu KPY. The Activation of the Mirror Neuron System during Action Observation and Action Execution with Mirror Visual Feedback in Stroke: A Systematic Review. Neural Plast. 2018 Apr 24;2018:2321045. doi: 10.1155/2018/2321045. eCollection 2018. PMID 29853839
- [Background] Gatti R, Rocca MA, Fumagalli S, Cattrysse E, Kerckhofs E, Falini A, Filippi M. The effect of action observation/execution on mirror neuron system recruitment: an fMRI study in healthy individuals. Brain Imaging Behav. 2017 Apr;11(2):565-576. doi: 10.1007/s11682-016-9536-3. PMID 27011016
- [Background] Wang J, Fritzsch C, Bernarding J, Holtze S, Mauritz KH, Brunetti M, Dohle C. A comparison of neural mechanisms in mirror therapy and movement observation therapy. J Rehabil Med. 2013 Apr;45(4):410-3. doi: 10.2340/16501977-1127. PMID 23474778
- [Background] Chen YH, Siow TY, Wang JY, Lin SY, Chao YH. Greater Cortical Activation and Motor Recovery Following Mirror Therapy Immediately after Peripheral Nerve Repair of the Forearm. Neuroscience. 2022 Jan 15;481:123-133. doi: 10.1016/j.neuroscience.2021.11.048. Epub 2021 Dec 5. PMID 34875363
- [Background] Thieme H, Morkisch N, Mehrholz J, Pohl M, Behrens J, Borgetto B, Dohle C. Mirror therapy for improving motor function after stroke. Cochrane Database Syst Rev. 2018 Jul 11;7(7):CD008449. doi: 10.1002/14651858.CD008449.pub3. PMID 29993119
- [Background] Willand MP, Rosa E, Michalski B, Zhang JJ, Gordon T, Fahnestock M, Borschel GH. Electrical muscle stimulation elevates intramuscular BDNF and GDNF mRNA following peripheral nerve injury and repair in rats. Neuroscience. 2016 Oct 15;334:93-104. doi: 10.1016/j.neuroscience.2016.07.040. Epub 2016 Jul 29. PMID 27476437
- [Background] Saavedra-Garcia A, Moral-Munoz JA, Lucena-Anton D. Mirror therapy simultaneously combined with electrical stimulation for upper limb motor function recovery after stroke: a systematic review and meta-analysis of randomized controlled trials. Clin Rehabil. 2021 Jan;35(1):39-50. doi: 10.1177/0269215520951935. Epub 2020 Aug 24. PMID 32830512
- [Background] Zhang Y, Zhang X, Cheng C, Huang S, Hua Y, Hu J, Wang Y, Zhang W, Yang Y, Liu Y, Jia J, Gou P, Zhang P, Zhou F, Wei X, Bai Y. Mirror therapy combined with contralaterally controlled functional electrical stimulation for the upper limb motor function after stroke: a randomized controlled trial. Disabil Rehabil. 2024 Jun;46(12):2528-2534. doi: 10.1080/09638288.2023.2225878. Epub 2023 Jun 21. PMID 37341447
- [Background] Loh MS, Kuan YC, Wu CW, Liao CD, Hong JP, Chen HC. Upper Extremity Contralaterally Controlled Functional Electrical Stimulation Versus Neuromuscular Electrical Stimulation in Post-Stroke Individuals: A Meta-Analysis of Randomized Controlled Trials. Neurorehabil Neural Repair. 2022 Jul;36(7):472-482. doi: 10.1177/15459683221092647. Epub 2022 May 16. PMID 35574940
- [Background] Huang JJ, Pei YC, Chen YY, Tseng SS, Hung JW. Bilateral Sensorimotor Cortical Communication Modulated by Multiple Hand Training in Stroke Participants: A Single Training Session Pilot Study. Bioengineering (Basel). 2022 Nov 24;9(12):727. doi: 10.3390/bioengineering9120727. PMID 36550934